CLINICAL TRIAL: NCT02745977
Title: Breast Milk Protein Intolerance and Maternal Dairy Consumption
Brief Title: Recruiting All Strictly Breast-fed Babies With Blood In Stool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Farrah Lazare, MD, Attending Physician, Pediatric Gastroenterology, Winthrop University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14021
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Breast Milk Protein Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dairy Free Diet- guaiac + on dairy free diet (Other): Dairy Free Diet x 3 weeks then stool guaiac positive
  Interventions: Other: Dairy Free Diet
- Guaiac negative on dairy free diet (Other): on dairy free diet x 3 weeks, then stool guaiac negative
  Interventions: Other: Dairy Free Diet

INTERVENTIONS:
Other: Dairy Free Diet — Dairy Free Diet x 3 stool guaiacs. If positive, dairy is reintroduced to diet.

SUMMARY:
Breast feeding is the most nutritious form of nourishment in infants and is recommended for at least the first four months of life. Breast fed infants may develop milk protein intolerance. The management of breast milk protein intolerance differs from that of cow's milk protein intolerance in formula fed infants. Because breast milk is considered by many to be nutritionally superior to formula and results in maternal infant bonding mothers are often told to continue breast feeding. Despite the lack of evidence based data to support or refute the modification of the mother's diet, it is suggested that they eliminate their own intake of dairy products strictly and avoid supplementing with a cow's milk based formula. Investigators are doing this study to demonstrate that the deletion of dairy from the diet of a breast feeding mother will not cause breast milk protein intolerance to resolve.

DETAILED DESCRIPTION:
Breast feeding is the most nutritious form of nourishment in infants and is recommended for at least the first four months of life. Breast fed infants may develop milk protein intolerance. The management of breast milk protein intolerance differs from that of cow's milk protein intolerance in formula fed infants. Because breast milk is considered by many to be nutritionally superior to formula and results in maternal infant bonding mothers are often told to continue breast feeding. Despite the lack of evidence based data to support or refute the modification of the mother's diet, it is suggested that they eliminate their own intake of dairy products strictly and avoid supplementing with a cow's milk based formula. The investigators are doing this study to demonstrate that the deletion of dairy from the diet of a breast feeding mother will not cause breast milk protein intolerance to resolve.Some infants have difficulty digesting breast milk. When this happens, the doctor may advise the mother to eliminate dairy from her diet as long as the mother continues breast feeding or until the baby is 12 months old. However, no studies have proven that this change in a mother's diet actually solves the baby's problem with breast milk. The purpose of this study is to find an answer to this question.

ELIGIBILITY:
Inclusion Criteria:

* Women with exclusively breast fed infants less than 4 months of age
* Infant that has a positive stool guaiac

Exclusion Criteria:

* Formula fed infants

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Presence of blood in the stool as evidenced by positive stool guaiac | 3 weeks
  If guaiac positive, then dairy is reintroduced to diet
guaiac negative on diary free diet | 3 weeks
  if guaiac negative on dairy free diet after 3 weeks, will rechallenge with dairy to prove that blood in stool is caused by dairy in mother's diet

CONTACTS AND LOCATIONS:
Locations (1):
- Winthrop Pediatric Associates, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: No